CLINICAL TRIAL: NCT04180995
Title: A Monocentric, Single-arm, Open, Phase II Clinical Study on the Efficacy and Safety of Toripalimab Combined With Axitinib as Neoadjuvant Therapy in Patients With Localized Mucosal Melanoma
Brief Title: Toripalimab in Combination With Axitinib in Patients With Localized Mucosal Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-132
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab, Axitinib (Experimental): The subjects will receive Toripalimab and Axitinib combined therapy after enrollment, and receive operation 2 weeks after the last dose of Axitinib. Toripalimab will be given for a total of 4 cycles (8 weeks), whereas Axitinib will be given for a total of 8 weeks.The subjects can receive Toripalimab for up to one year after the operation.
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 ) Axitinib tablet (Inlyta®)

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) Axitinib tablet (Inlyta®) — TORIPALIMAB INJECTION(JS001 ) combined with chemotherapy, 3mg/kg, Q2W,up to 1 years of treatment.

SUMMARY:
This study is one monocentric, single-arm, open, phase Ⅱ clinical study to evaluate the safety and efficacy of Toripalimab monoclonal injection (Tuo Yi) combined with axitinib tablet (Inlyta®) as neoadjuvant therapy for localized mucosal melanoma.

Primary objective: To evaluate pathological response (pCR+pPR) rate of Toripalimab combined with axitinib as neoadjuvant therapy for localized mucosal melanoma.

The subjects will receive Toripalimab and Axitinib combined therapy after enrollment, and receive operation 2 weeks after the last dose of Axitinib. Toripalimab will be given for a total of 4 cycles (8 weeks), whereas Axitinib will be given for a total of 8 weeks.The subjects can receive Toripalimab for up to one year after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Being voluntary to sign the informed consent form, with good compliance and willingness to cooperate with follow-up;
2. Age of 18-75 years, male or female;
3. Histopathologically diagnosed mucosal melanoma;
4. ECOG PS score 0 or 1;
5. Being considered to be able to be completely resected after multidisciplinary (including surgeon, oncologist and radiologist) discussion, and systemic staging examination improved prior to enrollment (need to include cranial enhanced CT/MRI, bone scan, thoracic, abdominal and pelvic enhanced CT/MRI (enhanced MRI of head and neck, gynecological examination additionally needed for female genital melanoma, colonoscopy additionally needed for rectal melanoma), B mode ultrasonography of superficial lymph node, or systemic PET-CT) demonstrated no regional or distant metastasis;
6. No contraindications for the treatment, including normal peripheral hemogram, basically normal hepatic and renal function as well as ECG:

   * Peripheral hemogram: white blood cell (WBC) ≥3.5×109/L, neutrophil (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (Hgb) ≥90 g/L;
   * Liver function: alanine aminotransferase (ALT) ≤1.5×ULN, aspartate aminotransferase (AST) ≤1.5×ULN, and total bilirubin (TBil) ≤1.5×ULN;
   * Renal function: blood urea nitrogen ≤ ULN, creatinine ≤ ULN;
7. Use of highly-effective contraceptive methods during the whole study for men of reproduction ability or women of pregnant possibility (e.g. oral contraceptives, intrauterine contraceptive device, abstinence of sexual intercourse or barrier contraception in combination with spermatocide), and continuation of contraception for 12 months after the end of study treatment.

Exclusion Criteria:

1. Previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2, or antiangiogenic drugs;
2. Known allergy to Toripalimab or Axitinib or excipient of the study drug;
3. Patients with ocular melanoma or melanoma with unknown primary foci;
4. Pregnant and breastfeeding women;
5. Abnormal coagulation function [activated partial thromboplastin time (APTT)> 43 s, or international normalized ratio (INR) > 1.5×ULN], or hemorrhagic tendency or hemorrhagic event occurred within two months prior to enrollment (e.g., gastrointestinal hemorrhage, hemorrhagic gastric ulcer, etc.), or receiving thrombolytic or anticoagulation therapy;
6. Currently having serious and uncontrolled acute infection, or suppurative infection, chronic infection, or prolonged wound healing;
7. Having serious heart disease, including congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, severe valvular heart disease and refractory hypertension;
8. Having neurological, mental disease or psychiatric disorder that can not be easily controlled, poor compliance, inability to cooperate and narrate therapeutic response;
9. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
10. Concomitantly other Malignancies;
11. Concomitant participation in other clinical trials;
12. Positive HIV antibody, or positive HCV antibody/HCV-RNA, or positive HBsAg or HBcAb whilst HBV DNA copy >2000 IU/ml;
13. Active autoimmune diseases requiring systemic treatment in the past two years (e.g., use of disease-regulating drug, corticosteroid or immunosuppressant), relevant replacement therapy is allowed (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency);
14. Vaccination of live vaccine within 4 weeks prior to the start of study;
15. Other severe, acute or chronic medical diseases or abnormalities in laboratory examination possibly increasing the relevant risk in study participation or possibly interfering the interpretation of study results as judged by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-07-06 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological response (pCR+pPR) rate: defined as the percentage of subjects without alive tumor cells and alive tumor cells in postoperative resected specimens 10% - 50% in the resected specimen post operation. | Approximately 8 weeks
  To evaluate pathological response (pCR+pPR) rate of Toripalimab combined with axitinib as neoadjuvant therapy for localized mucosal melanoma.

SECONDARY OUTCOMES:
RFS (recurrence-free survival) per RECIST1.1 as Assessed by investigator | Approximately 1 years
  To evaluate recurrence-free survival (RFS) of Toripalimab combined with axitinib as neoadjuvant therapy for localized mucosal melanoma.
OS (overall survival) | Approximately 2 years
  OS at 1 or 2 years.
Incidence of AEs/SAEs | Approximately 2 years
  Adverse events (AEs) ; serious adverse events (SAEs); abnormal value of Lab test according to NCI-CTCAE V5.0
Pathological complete response (pCR) rate: defined as the percentage of subjects without alive tumor cells in the resected specimen post operation. | Approximately 8 weeks
  To evaluate pathological complete response (pCR) rate of Toripalimab combined with axitinib as neoadjuvant therapy for localized mucosal melanoma.

OTHER OUTCOMES:
PD-L1 expression | 2 years
  Correlation between predictive biomarkers and efficacy, including PD-L1 expression.
CD3 and CD8 gene mutation | 2 years
  Correlation between predictive biomarkers and efficacy, including CD3 and CD8, gene mutation status, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China